CLINICAL TRIAL: NCT06943170
Title: Effects of Aerobic Exercise With and Without Low Calorie Diet on Adiposity and BMI of Overweight and Obese Children With Down Syndrome
Brief Title: Aerobic Exercise With and Without Low Calorie Diet on Adiposity and BMI of Down Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR/AHS/24/0722
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Down Syndrome
Keywords: Down Syndrome, Obesity, Adiposity, Body Mass Index (BMI)
MeSH Terms: conditions — Down Syndrome; Obesity | interventions — Exercise; Caloric Restriction

STUDY DESIGN:
Intervention Model Description: * Experimental Group I: Aerobic Exercise with Low Calorie Diet.
  * Experimental Group II: Aerobic Exercise without Low Calorie Diet.
  FITT Principle The exercise groups will follow a supervised 12-week aerobic training intervention program. The duration of each aerobic exercise session will be set at 10 min for the first two weeks, 20 min for the next two weeks, and 30 min for the remaining eight weeks.
  Brisk Walk, a type of moderate intensity aerobic exercise can be an effective component of a weight loss program for overweight and obese children with Down syndrome.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group and the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise With Low Calorie Diet (Experimental): EXPERIMENTAL GROUP I Detailed FITT Protocol of Aerobic Exercise
  Warm-Up Exercise Cool-Down
  Low Calorie Diet Plan:
  Intermittent Fasting (12 hours for first 4 weeks and 16 hours for remaining 8 weeks)
  Interventions: Other: Aerobic Exercise and Low Calorie Diet
- Aerobic Exercise without low calorie diet (Experimental): Warm Up Exercise Cool down
  Interventions: Other: Aerobic Exercise and Low Calorie Diet

INTERVENTIONS:
Other: Aerobic Exercise and Low Calorie Diet — Group A: Aerobic Exercise with Low calorie diet Group B: Aerobic Exercise without Low Calorie Diet

SUMMARY:
Down syndrome (DS) is caused by trisomy 21, or the presence of an extra copy of chromosome 21. A calibrated weight scale is used to measure participants' weight accurately. A stadiometer measures participants' height to the nearest millimeter. A flexible non-stretchable waist circumference tape is used to assess abdominal obesity. Body mass index (BMI, ratio of height and weight, expressed as kg/m2 6-Min Walk is a test to evaluate aerobic fitness level. Brisk Walk, a type of moderate intensity aerobic exercise can be an effective component of a weight loss program for overweight and obese children with Down syndrome. The aim of this study to compare the effects of aerobic exercise alone versus aerobic exercise combined with a low calorie diet, to provide insights into optimal inte A randomized controlled trial will be conducted. The study will be conducted at Rehab Clinic, Lahore in a total duration of 10 months. Sample size will be 22. There will be two study groups, Group I: Aerobic Exercise with Low calorie diet and Group II: Aerobic Exercise without Low calorie diet. Non-Probability Convenient sampling technique will be used to collect the data.

DETAILED DESCRIPTION:
Down syndrome (DS) is caused by trisomy 21, or the presence of an extra copy of chromosome 21. About 1 in 800 newborns globally experience it. The unusual phenotype that characterizes children with DS is thought to be caused by an overabundance of chromosome 21 genes or a breakdown of genetic balance. Up slanting palpebral fissures, epicanthic folds, and brachycephaly are nearly universal features of Down syndrome. Obstetricians have adopted a new paradigm for Down syndrome screening. Combined overweight and obesity prevalence was 23-70% (overweight: 13.3-52.9%; obesity: 0-62.5%). Interventions for obesity prevention and control are primarily based on diet and exercise-based programs. A calibrated weight scale is used to measure participants' weight accurately. A stadiometer measures participants' height to the nearest millimeter. A flexible non-stretchable waist circumference tape is used to assess abdominal obesity. Body mass index (BMI, ratio of height and weight, expressed as kg/m2 6-Min Walk is a test to evaluate aerobic fitness level. Brisk Walk, a type of moderate intensity aerobic exercise can be an effective component of a weight loss program for overweight and obese children with Down syndrome. The aim of this study to compare the effects of aerobic exercise alone versus aerobic exercise combined with a low calorie diet, to provide insights into optimal interventions for reducing adiposity and improving BMI in this vulnerable population.

A randomized controlled trial will be conducted. The study will be conducted at Ghurki Trust and Teaching Hospital (GTTH) and Rehab Clinic, Lahore in a total duration of 10 months. Sample size will be 22. There will be two study groups, Group I: Aerobic Exercise with Low calorie diet and Group II: Aerobic Exercise without Low calorie diet. Non-Probability Convenient sampling technique will be used to collect the data. The Following sample characteristics will be included in the study: Children with diagnosed Down Syndrome, age (8-14 years), Both Genders (male and female), BMI (85TH-95TH percentile), generally stable health condition with parents' approval to participate in the study. The population having the following characteristics will be excluded from the study: History of any previous medical disease, previous participation in any Weight Loss Exercise Program or any specific diet plan from last 6 months, children on medication that could affect weight or metabolism, children with physical disabilities and cognitive impairments and with dietary restrictions or food allergies. The tools that will be included in the study are: Digital Weight Scale, Stadiometer, BMI calculator, Skin-Fold Caliper, 6 min walk test, rate of perceived exertion (RPE) Scale and Food Frequency Questionaire. Aerobic Exercise and Low calorie diet will be used as intervention. SPSS version 27 will be used for data analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age (8-16) years.
* Both Genders (Male and Female).
* BMI-for-age percentile (at or above 85th percentile is overweight, and at or above 95th percentile is considered as obese)
* Children with generally stable health condition, without significant co-morbidities that might affect diet or exercise interventions.
* Consent form signed by parents, along with written approval by the physician.

Exclusion Criteria:

* History of any previous medical disease.
* Previous Participation in any Weight Loss Exercise Program.
* Participants following any specific diet plan from last 6 months.
* Exclusion of children on medication that could affect weight or metabolism.
* Children with physical disabilities that prevent them from safely participating in aerobic exercise.
* Children with dietary restrictions or food allergies.
* Children with severe cognitive impairments that prevent them from engaging in exercise program.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Digital weight Scale | Baseline and 12th week
  A calibrated scale is used to measure participants' weight accurately. It should be placed on a level surface and calibrated regularly to ensure precision.
  2. S A calibrated scale is used to measure participants' weight accurately. It should be placed on a level surface and calibrated regularly to ensure precision.
  2. S Tool to measure participant's weight accurately.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Baseline and 12th week
  To measure particpants adiposity

OTHER OUTCOMES:
Waist Circumference Measurements | baseline and 12th week
  To measure abdominal adiposity
Skin Fold thickness | Baseline and 12th week
  To measure skin fold thickness at various anatomical points

CONTACTS AND LOCATIONS:
Overall Officials: Jannat Arshad, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- Jannat Arshad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antonarakis SE, Skotko BG, Rafii MS, Strydom A, Pape SE, Bianchi DW, Sherman SL, Reeves RH. Down syndrome. Nat Rev Dis Primers. 2020 Feb 6;6(1):9. doi: 10.1038/s41572-019-0143-7. PMID 32029743
- [Background] Bull MJ. Down Syndrome. N Engl J Med. 2020 Jun 11;382(24):2344-2352. doi: 10.1056/NEJMra1706537. No abstract available. PMID 32521135
- [Background] Ergaz-Shaltiel Z, Engel O, Erlichman I, Naveh Y, Schimmel MS, Tenenbaum A. Neonatal characteristics and perinatal complications in neonates with Down syndrome. Am J Med Genet A. 2017 May;173(5):1279-1286. doi: 10.1002/ajmg.a.38165. Epub 2017 Apr 6. PMID 28386951
- [Background] Saghazadeh A, Mahmoudi M, Dehghani Ashkezari A, Oliaie Rezaie N, Rezaei N. Systematic review and meta-analysis shows a specific micronutrient profile in people with Down Syndrome: Lower blood calcium, selenium and zinc, higher red blood cell copper and zinc, and higher salivary calcium and sodium. PLoS One. 2017 Apr 19;12(4):e0175437. doi: 10.1371/journal.pone.0175437. eCollection 2017. PMID 28422987
- [Background] Krivega M, Stiefel CM, Storchova Z. Consequences of chromosome gain: A new view on trisomy syndromes. Am J Hum Genet. 2022 Dec 1;109(12):2126-2140. doi: 10.1016/j.ajhg.2022.10.014. PMID 36459979
- [Background] Gonzalez-Aguero A, Vicente-Rodriguez G, Moreno LA, Guerra-Balic M, Ara I, Casajus JA. Health-related physical fitness in children and adolescents with Down syndrome and response to training. Scand J Med Sci Sports. 2010 Oct;20(5):716-24. doi: 10.1111/j.1600-0838.2010.01120.x. PMID 20456681